CLINICAL TRIAL: NCT02587130
Title: The Effect and Tolerance of a Ketamine Subcutaneous Bolus, During Painful Care of Refractory Bed Sores, Ulcers and Vascular Wounds in a Palliative Care Unit
Brief Title: Ketamine and Refractory Painful Care in a Palliative Unit
Acronym: KETAREF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: difficulted recruiting
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC-P0041
Record Dates: First submitted 2015-10-13; First posted 2015-10-27 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Intractable Pain; Intensive Care; Pressure Ulcer; Pain Management
Keywords: intractable pain; pressure ulcer; bed sore; palliative medicine; ketamine; pain management
MeSH Terms: conditions — Pain, Intractable; Pressure Ulcer; Agnosia | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- communicating and none-communicating patients (Experimental): 20 communicating patients (evaluated with the visual analogue pain scale (VAS)) and 20 none-communicating patients or patients presenting cognitive disturbance or vigilance (evaluated with the Algoplus scale)
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — ketamine administered in bolus by subcutaneous injection

SUMMARY:
Pain is one of the major symptoms in palliative care units and often is very difficult to treat, being considered as a refractory pain.

There are different causes of refractory pain: pain due to bed sores and ulcer bandages, carcinological or ischemic wounds or injuries, pain due to patients' reduced mobility, pain due to traumatological injuries, pain associated with a long-term bed confinement, etc.

The investigators propose a prospective study to estimate the effect and the tolerance to a subcutaneous bolus of ketamine administered for the treatment of refractory pain due to the care of bedsores, ulcers and vascular wounds in patients hospitalized in palliative care units.

DETAILED DESCRIPTION:
Patients in palliative care units have serious and incurable conditions and are in the sickness' late or final stages. This is why the relief of their symptoms is a priority for their medical care, being pain one of the major symptoms.

In this context, the idea of treating various types of pain such as pain due to bed sore and ulcer bandages, carcinological or ischemic wounds or injuries, pain due to patients' reduced mobility, etc. was raised.

French Ministry of Health's 2010 recommends the use of ketamine to treat refractory pain after the failure of usual therapeutic treatments (opioids, Nitrous oxide and oxygen (also known as MEOPA)). This treatment is then used in association with midazolam (0.01 to 0.05 mg/kg) to prevent hallucinating effects.

However, the intravenous treatment is often the alternative and this choice is justified by the study population's characteristics (usually elderly patients, multi-pathologic, etc) and by the invasive way of treatment used with a repeated central and peripheral venous catheters which is contrary to the primary objective of patient comfort.

To the investigators' knowledge, no randomised study has ever been done regarding the use of ketamine to treat refractory pain administered subcutaneously.

ELIGIBILITY:
Inclusion Criteria:

* Patients of ≥18 years old, hospitalized in palliative care units
* Conscious or presenting altered/disturbed consciousness but for whom the Rudkin score is ≤ 4 (eyes closed, response to light tactical stimulation)
* For whom a palliative care is acted
* No matter the progression and prognostic status
* After the information is given to the patient (with the notification form given) and the written consent form is retrieved and when the state of cognition and vigilance allows it. In case of cognitive and consciousness disturbance, after informing and retrieving the written consent form from the patient's trusted person, or a relative by default, for patients under guardianship after being informed and giving a consent form written by the legal representative.
* Evened out on an analgesia level, without care
* Who has not received ketamine for 60 days before inclusion no matter the indications
* For whom bedsore, ulcer or vascular injuries have appeared and continue to be painful despite the administration of opioid bolus with the painful evaluation regarding the visual analogic scale (EVA) ≥ 5/10, or regarding the evaluation of the Algoplus pain behavior scale ≥ 2, or for whom the opioid treatment cannot be administered due to the presence of adverse side effects (drowsiness, confusion, nausea, vomiting, respiratory depression…)
* And for whom caring under Entonox (a medical analgesic gas which is a mix of nitrous oxide and oxygen) is inefficient or not compatible.
* Lack of easy venous access

Exclusion Criteria:

* Contraindication of Ketamine in case of anesthesia (AMM) : allergy, porphyria
* Late stage heart failure
* Intracranial hypertension
* Acute heart attack phase
* Unstable psychosis
* Presence of agitation
* Pregnant woman
* Patient with no affiliation to a social security system
* Contraindication of Midazolam: known hypersensitivity to benzodiazepines or any other know excipient of the product, acute respiratory depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Pain Score on the Visual Analog Scale or Algoplus after subcutaneous bolus of Ketamine | 2 hours
  Evaluate the symptomatic effect on pain and the comfort of ketamine's sub-cutaneous bolus administered to adults hospitalized in palliative units during painful care of vascular wounds, ulcers and bedsores, not eased by opioid or Entonox (a medical analgesic gas which is a mix of nitrous oxide and oxygen) or for whom these treatments are not adapted (Entonox, in cases of disturbed consciousness) or for whom side effects are unbearable (drowsiness, confusion, nausea, vomiting, respiratory depression…). Two kind of scores will be analyzed (EVA and Algoplus).

SECONDARY OUTCOMES:
Number of secondary side effects after administration of a sub-cutaneous ketamine's bolus | 2 hours
  Evaluate the tolerance of the sub-cutaneous administration of ketamine's bolus, with protocol dosages and with the surveillance of:
  * Arterial pressure, heart frequency, respiratory frequency, saturation in visual oxygen
  * The appearance of neuroleptic symptoms: confusion, perturbation of visual/hearing sensations, humor perturbation, hallucinations, agitation…
  * Appearance of hypersialorrhea, bronchial cluttering
  * Presence of nausea or vomiting
  * Presence of cephalgia or dizziness
Ketamine dosage administered in sub-cutaneous bolus before painful caring | 2 hours
  Define a ketamine dosage administered in sub-cutaneous bolus, before painful caring in order to obtain the antalgic efficacy thanks to EVA < 3 or Algoplus scale < 2, and in a satisfactory efficacy/tolerance report for patients' comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Danel Delerue, MD, Principal Investigator — Groupment des Hôpitaux de l'Institut Catholique de Lille
Locations (1):
- GHICL, Lomme, France